CLINICAL TRIAL: NCT01837654
Title: Plantarflexion Reduces Urgency and Peak Detrusor Pressure in Patients With Detrusor Overactivity
Acronym: DO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 76/12
Record Dates: First submitted 2013-04-18; First posted 2013-04-23 (Estimated); Results first posted 2019-03-11 (Actual); Last update posted 2019-03-11 (Actual); Status verified 2018-11

CONDITIONS: Overactive Detrusor
Keywords: Detrusor Overactivity; Plantarflexion; Urgency
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Plantarflexion - 2nd wave (Experimental): At the beginning of the 2nd wave, patients will be asked to perform continuous plantar-flexion by pushing their tiptoes against the floor.
  Interventions: Behavioral: Plantarflexion 2nd wave
- Plantarflexion - 3rd wave (Experimental): At the beginning of the 3rd wave, patients will be asked to perform continuous plantar-flexion by pushing their tiptoes against the floor.
  Interventions: Behavioral: Plantarflexion - 3rd wave

INTERVENTIONS:
Behavioral: Plantarflexion 2nd wave — At the beginning of the 2nd wave, patients will be asked to perform continuous plantar-flexion by pushing their tiptoes against the floor.
  Arms: Plantarflexion - 2nd wave
Behavioral: Plantarflexion - 3rd wave — At the beginning of the 3rd wave, patients will be asked to perform continuous plantar-flexion by pushing their tiptoes against the floor.
  Arms: Plantarflexion - 3rd wave

SUMMARY:
The purpose of this study is to find out whether plantarflexion has an effect on the degree of urinary urgency and on the amplitude of detrusor contraction during filling cystometry in patients with detrusor overactivity (DO).

DETAILED DESCRIPTION:
Patients with urodynamic DO will be included in this study. During urodynamics, the mean peak detrusor pressures of each contraction will be documented and compared. At the beginning of the 2nd or 3rd wave, patients will be asked to perform continuous plantar-flexion by pushing their tiptoes against the floor. Following each wave, patients will be asked to grade the severity of the urgency by a visual analogue scale

ELIGIBILITY:
Inclusion Criteria:

All patients with urodynamic detrusor overactivity

Exclusion Criteria:

Inability to perform plantarflexion due to mental or physical disability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2012-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kobi Stav, MD, Principal Investigator — Assaf Harofe Medical Center
Locations (1):
- Assaf Harofe Medical Center, Be’er Ya‘aqov, Israel

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Ninety three consecutive patients underwent multichannel urodynamic study. All patients were referred for urodynamics in order to evaluate lower urinary tract symptoms. Twenty seven were diagnosed with DO. Twenty two patients were included in the study and comprised the study cohort. Five patients were excluded due to physical disability.
Pre-assignment Details: Twenty seven patients were diagnosed with DO. Twenty two patients were included in the study and comprised the study cohort. Five patients were excluded due to physical disability.
Groups:
- Plantarflexion - 2nd Wave of Contraction: At the beginning of the 2nd wave, patients will be asked to perform continuous plantar-flexion by pushing their tiptoes against the floor.
  Plantarflexion 2nd wave : At the beginning of the 2nd wave, patients will be asked to perform continuous plantar-flexion by pushing their tiptoes against the floor.
- Plantarflexion - 3rd Wave of Contraction: At the beginning of the 3rd wave, patients will be asked to perform continuous plantar-flexion by pushing their tiptoes against the floor.
  Plantarflexion - 3rd wave : At the beginning of the 3rd wave, patients will be asked to perform continuous plantar-flexion by pushing their tiptoes against the floor.
Period: Overall Study
Arm/Group | Plantarflexion - 2nd Wave of Contraction | Plantarflexion - 3rd Wave of Contraction
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Plantarflexion - 2nd Wave: At the beginning of the 2nd wave, patients will be asked to perform continuous plantar-flexion by pushing their tiptoes against the floor.
  Plantarflexion 2nd wave : At the beginning of the 2nd wave, patients will be asked to perform continuous plantar-flexion by pushing their tiptoes against the floor.
- Plantarflexion - 3rd Wave: At the beginning of the 3rd wave, patients will be asked to perform continuous plantar-flexion by pushing their tiptoes against the floor.
  Plantarflexion - 3rd wave : At the beginning of the 3rd wave, patients will be asked to perform continuous plantar-flexion by pushing their tiptoes against the floor.
- Total: Total of all reporting groups
Arm/Group | Plantarflexion - 2nd Wave | Plantarflexion - 3rd Wave | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 8
  >=65 years | 7 | 7 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (11) | 68 (12) | 67 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 6 | 6 | 12
Region of Enrollment [Number; unit: participants]
  Israel | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Mean Peak Detrusor Pressures
Description: Mean peak detrusor pressures of each contraction
Time Frame: through test completion, an average of 10 minutes
Measure: Mean (Standard Deviation); unit: cm H2O
Arm/Group | Plantarflexion - 2nd Wave | Plantarflexion - 3rd Wave
Number analyzed (Participants) | 11 | 11
cm H2O | 58 (14) | 31 (19)

2. Secondary Outcome: Severity of the Urgency by a 0-10 Visual Analogue Scale (VAS).
Description: Following each wave, patients will be asked to grade the severity of the urgency by a 0 (minimum) to 10 (maximum) visual analogue scale (VAS).
Time Frame: through test completion, an average of 10 minutes
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Plantarflexion - 2nd Wave | Plantarflexion - 3rd Wave
Number analyzed (Participants) | 11 | 11
units on a scale | 4.7 (1.8) | 4.7 (1.7)

ADVERSE EVENTS:
Arm/Group | Plantarflexion - 2nd Wave | Plantarflexion - 3rd Wave
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes